CLINICAL TRIAL: NCT06823492
Title: Effects of Early Trauma on Neurocognitive Development and Mental Health
Brief Title: Investigating the Impacts of Early Life Experience on the Brain & Behaviour
Status: Recruiting | Type: Observational
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Rebecca Elliot, Prof Chair in Affective Neuroscience, University of Manchester
Other Study IDs: 2024-17962-32800
Record Dates: First submitted 2024-12-10; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Mental Health; Neurodevelopment; ADHD; Autism; Depression - Major Depressive Disorder; Anxiety Disorder (Panic Disorder or GAD)
Keywords: fMRI; cognition; brain imaging; adoption; trauma
MeSH Terms: conditions — Psychological Well-Being; Attention Deficit Disorder with Hyperactivity; Autistic Disorder; Anxiety Disorders; Panic Disorder; Generalized Anxiety Disorder; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control Group: Young adults, aged 18-15 who were not adopted and have no experience of childhood trauma
- Adopted Group: Young adults, aged 18-15 who were adopted

SUMMARY:
The aim of this study is to learn more about how early life experience influences the brain, behaviour, and the immune system later in life. This will help improve understanding of why certain early life experiences (e.g., adoption, stress and parental separation) can cause difficulties for some people when they are adults. The long-term goal of this research is to develop tools that could identify young people who are vulnerable to developing future problems, this will ensure people get the help that they need at the right time for them.

This study will use psychological assessment, online games, brain imaging and blood sampling to help improve our understanding of how and why early life experience can influence mental health, cognition, brain development and the immune system later in life.

DETAILED DESCRIPTION:
Step 1: Telephone/Video screening call (20 minutes)

The first part of this study is a brief telephone/video call during which you will:

* Be asked questions to check whether you meet the study eligibility criteria.
* Be asked questions about your medical history (including mental health) and use of psychiatric medication.

Step 2: ONLINE PARTS OF THE STUDY (3 hours) Once you have completed the online consent form you will be emailed a link to the online parts of the study.

* You will be asked to fill in three online questionnaires which take around 30 minutes each and collect information about your demographics (e.g., sex, job, ethnicity, income etc.,), medical history, mental health conditions (e.g., autism spectrum quotient (you may opt of this questionnaire), depression, anxiety, addiction, drug and alcohol use) and personality traits (e.g., impulsivity, attachment, neuroticism, extraversion).
* You will be asked to complete online games which are designed to assess memory, impulsivity, attention, face recognition and social interaction. These short tasks (5 - 10 minutes each) are similar to simple "brain training" games you may have seen online. They will take around 1.5 hours to complete in total.

Step 3: FACE-TO-FACE PARTS OF THE STUDY (2-hours)

BRAIN SCAN (1.5 hours)

* When you arrive, you will be asked to review this study information sheet and sign a paper consent form and other safety/screening forms required for the study.
* You will then be asked to take part in a magnetic resonance imaging (MRI) brain scan. You will be asked to lie down in a strong magnetic field for an hour whilst a computer takes pictures of your brain, and you complete short cognitive tasks (3 x 10 minutes each) and a resting state brain scan (10 minutes).

BLOOD TEST (30 minutes) We would also like to collect a blood sample from you, as this will help us understand how early life events can impact your white blood cells which are a key part of your immune system.

Step 4: INTERVIEWS, QUESTIONNAIRES & MEMORY GAME (1.5 - 3 hours)

You can choose to do the following parts of the study either when you visit the University of Manchester or during a remote session (Zoom/telephone).

* The researcher will conduct interviews about your mental health history and your experience of friendships and relationships (up 2.5 hours).
* You will be asked to complete a short, anonymised questionnaires about your experience of trauma and stress in your childhood including the Childhood Trauma Questionnaire and the Adverse Childhood Experiences questionnaire (15 minutes).
* You will complete a short emotional memory game (on the researchers' laptop or via your computer if via Zoom) (5 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-24
* Reside in Greater Manchester
* You are not enrolled on a university degree course and do not hold a university degree qualification
* Lived with one or both birth parents throughout childhood.
* Able to travel to the University of Manchester
* Able to understand the study information and participate in the assessment procedures described below (independently or with reading support from a researcher, friend or family member)
* Able to read text on a computer screen (using glasses or contact lenses if required)
* To sign up for this study one or more of the following statements should apply to you:

  1. I am not currently in education employment or training, or I am unemployed.
  2. I receive benefits from the Government e.g., housing benefits, universal credit, personal independent payment (PIP), disability benefit, job seekers allowance.
  3. I am currently struggling due mental health problems or neurodiversity (e.g., depression, anxiety, ADHD, autism, eating disorder)

Exclusion Criteria:

* You were looked after by the local authority (e.g., foster, kinship care or residential children's home) or adopted during childhood.
* Any experience of childhood trauma (including neglect, physical/verbal abuse, sexual abuse or exposure to domestic violence).
* Your family required input from social services due to child protection concerns.
* You are experiencing symptoms of and have been diagnosed with Post-Traumatic Stress Disorder (PTSD), borderline personality disorder (BPD), Emotionally Unstable Personality Disorder (EUPD).

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Control Group (Non-Adopted)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Mental health prevalence | January 2027
  Will be assessed on an individual subject level using the Structured Clinical Interview for DSM-V (SCID-5). (Outcome Measure: Summary counts of participants in each group showing the occurrence of different mental health disorders)
Neurodevelopmental condition prevalence | March 2027
  Autism will be assessed using the online screening tool, Autism Spectrum Quotient (ASQ) and the Autism Diagnostic Observation Schedule (ADOS). (Outcome Measure: Summary counts of participants in each group showing the occurrence of different neurodevelopmental disorders)
Neural Processing Differences related to childhood trauma and mental health: whole brain anlaysis | March 2027
  fMRI analyses will first be analysed using a typical univariate approach using Statistical Parametric Mapping. Exploratory whole brain analyses will be conducted. Statistical comparisons will be made between the adopted and control groups.
  Outcome measure: BOLD signal change in brain regions identified during whole brain comparisons which are associated with specific conditions of interest/task contrasts, and how these differ between the groups.

SECONDARY OUTCOMES:
Employment | March 2027
  This data will be collected using self-report online questionnaires. (Outcome Measure: Summary counts of participants in each group showing the occurrence of different levels of employment)
Education level | March 2027
  This data will be collected using self-report online questionnaires. (Outcome Measure: Summary counts of participants in each group showing the occurrence of different levels of education)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Biology Medicine & Health, University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No